CLINICAL TRIAL: NCT03156647
Title: Alpha-synuclein Level in the Saliva as a Potential Diagnostic Aid to Differentiate Between Idiopathic Parkinson Disease and Iatrogenic Parkinsonian Syndrome
Brief Title: Alpha-synuclein Level in Saliva to Differentiate Between Idiopathic Parkinson Disease and Iatrogenic Parkinsonian Syndrome
Acronym: PARKSYN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2016/GC-01bis
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Parkinson Disease; Parkinsonian Disorders
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- idiopathic Parkinson disease
  Interventions: Diagnostic Test: Level of alpha-synuclein
- iatrogenic parkinsonian syndrome
  Interventions: Diagnostic Test: Level of alpha-synuclein
- healthy volunteers
  Interventions: Diagnostic Test: Level of alpha-synuclein

INTERVENTIONS:
Diagnostic Test: Level of alpha-synuclein — Test of levels of total and ratio total:oligomeric in saliva

SUMMARY:
The aim of this study is to determine whether a significant reduction in the total level of alpha-synuclein and significant increase in the oligomeric form of alpha-synuclein and therefore the ratio oligomeric:total alpha-synuclein occurs in patients with Parkinson disease compared to patients with drug-induced parkinsonian syndrome.

ELIGIBILITY:
Inclusion Criteria

* The patient must have given their free and informed consent and signed the consent form
* The patient must be insured or the beneficiary of an insurance policy
* The patient is less than 55 years old
* For patients with acquired parkinsonian syndrome (UKPDSBB criteria) currently at HOEHN and YAHR stage ≤3:

  * For patients recruited via a psychiatrist: after anti-dopamine treatment
  * For patients recruited via a neurologist: having a recent diagnosis (≤2 years) of Parkinson disease

Exclusion Criteria:

* The subject is participating in another study
* The subject is in an exclusion period determined by a previous study
* The patients is under judicial protection
* The subject or their representative refused to sign the consent form
* It proves impossible to give the subject or their representative clear information.
* Patients with atypical degenerative parkinsonian syndrome
* Patients with vascular, post-traumatic, metabolic, toxic or genetic parkinsonian syndrome
* Appearance of parkinsonian syndrome prior to treatment with anti-dopamine
* Injection of botulinum toxin into the salivary glands
* Contra-indication on DAT-scan (unbalanced dysthyroidism, allergy, treatment with bupropion or amphetaminergics)
* Poor oral health (polyposis, gingivostomatitis) observed during the odontologist visit
* Patients not taking anti-psychotics with parkinsonian syndrome and normal DAT-scan

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Subjects will be recruited from three centres:
  Patients hospitalized in the Quissac psychiatric unit Patients followed in the CHU Nimes neurological department for idiopathic Parkinson Patients followed in the CHU Montpellier neurological department
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Compare saliva level of oligomeric alpha-synuclein between two groups of patients wth classical parkinsonian: patients with idiopathic Parkinson disease and patients with a acquired parkinsonian syndrome from anti-dopamine treatment. | Day 0

SECONDARY OUTCOMES:
Perform the first estimation of discriminatory capacity of saliva levels of oligomeric alpha-synuclein for diagnostic differentiation between idiopathic Parkinson disease and anti-dopamine induced acquired parkinsonian syndrome. | Day 0
Compare levels of total alpha-synuclein and the ratio of oligomeric alpha-synuclein:total alpha-synuclein between the two groups | Day 0
Perform the first estimation of discriminatory capacity of saliva levels of total oligomeric alpha-synuclein and the ratio of oligomeric alpha-synuclein:total alpha-synuclein for diagnostic differentiation between two groups | Day 0
Creation of a biobank with remaining samples | Day 0
  saliva samples
UPDRS II-III-IV score | Day 0
UDysRs score | Day 0
character of parkinsonian syndrome | Day 0
  symmetrical or asymmetrical
akathisia | Day 0
questionnaire on non-motor symptoms in Parkinson disease | Day 0
  PD-NMS
neuro-psychological evaluation | Day 0
  BREF+MOCO score
GDS score | Day 0
interogation to determine extent of motor and non-motor clinical markers to differentiate the two groups | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Castelnovo, MD, Principal Investigator — CHU Nimes
Locations (3):
- France (3):
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital St Eloi, Montpellier
  - CHU Nimes, Nîmes

IPD SHARING:
Plan to Share IPD: No